CLINICAL TRIAL: NCT03246724
Title: A Single-center, Randomized, Double-blind, Double-dummy, Parallel-group Study Comparing Oral Sedation to Intravenous Sedation for Ocular Procedures.
Brief Title: Oral Versus Intravenous Sedation for Ocular Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: H-36590
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Surgery; Sedation
Keywords: Ocular surgery; Intravenous sedation; Oral sedation
MeSH Terms: interventions — Triazolam; Midazolam; microcrystalline cellulose; Cellulose; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Interventions: triazolam oral sedation with sodium chloride 0.9% IV placebo or microcrystalline cellulose oral placebo with midazolam IV sedation
  Subjects will be randomized (1:1) to one of the two study arms listed above. On the day of surgery, the subject, anesthesiologist/CRNA, and surgeon will be blinded to the treatment assignment. The anesthesiologist/CRNA or pre-operative nurses will administer the blinded oral medication approximately 30 minutes before the procedure beings. The anesthesiologist/CRNA will administer the blinded IV medication approximately 5 minutes before the procedure begins. At the completion of the procedure, the anesthesiologist/CRNA and the surgeon will complete a satisfaction survey. The subject will then return within 2 days for their first post-operative clinical visit and complete a satisfaction survey.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subject and their entire medical team (including the anesthesiologist and surgeon) will all be masked to the subject's randomized intervention group. The randomization groups will be assigned by the statistician who will be unmasked. All medications will be provided to the medical team on the day of the procedure completely masked. The clinical research coordinator, the clinical research assistant, and the pharmacy will be unmasked to the intervention group. Any member of the medical team can be unmasked at any time after the intervention is administered in the case of an emergency resulting in a serious adverse event or an unanticipated problem.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cataract Procedures (Experimental): The following ocular procedures will fall under this arm of the study:
  • Cataracts
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Interventions: Drug: Triazolam; Drug: Midazolam; Drug: Microcrystalline Cellulose; Drug: Sodium chloride 0.9%
- Retina Procedures (Experimental): The following ocular procedures will fall under this arm of the study:
  * Pars plana vitrectomy
  * Pars plana vitrectomy with cataracts, epiretinal membrane peel, pars plana lensectomy, and/or endolaser, silicone oil removal
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Interventions: Drug: Triazolam; Drug: Midazolam; Drug: Microcrystalline Cellulose; Drug: Sodium chloride 0.9%
- Cornea Procedures (Experimental): The following ocular procedures will fall under this arm of the study:
  * Descemet Stripping Endothelial Keratoplasty (DSEK)
  * Cataracts with Descemet Stripping Endothelial Keratoplasty (DSEK)
  * Descemet Membrane Endothelial Keratoplasty (DMEK)
  * Cataracts with Descemet Membrane Endothelial Keratoplasty (DMEK)
  * Conjunctival and/or corneal lesion excisions
  * Pterygium
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Interventions: Drug: Triazolam; Drug: Midazolam; Drug: Microcrystalline Cellulose; Drug: Sodium chloride 0.9%
- Glaucoma Procedures (Experimental): The following ocular procedures will fall under this arm of the study:
  * Ahmed valve
  * Ahmed valve with cataracts
  * Trabeculectomy
  * Trabeculectomy with cataracts
  * Baerveldt
  * Baerveldt with cataracts
  * Endocyclophotocoagulation
  * Endocyclophotocoagulation with cataracts
  * Istent
  * Cataracts with istent
  * Kahook
  * Cataracts with kahook
  * Cypass
  * Cypass with cataracts
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Interventions: Drug: Triazolam; Drug: Midazolam; Drug: Microcrystalline Cellulose; Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Triazolam — This will be used for oral sedation. This capsule or a microcrystalline cellulose placebo capsule will be administered depending on the randomized treatment group.
  Dose for BMI less than 35: 0.125 mg
  Dose for BMI greater than or equal to 35: 0.25 mg
  Other Names: Halcion
Drug: Midazolam — This will be used for intravenous sedation. This injection or sodium chloride 0.9% will be administered depending on the randomized treatment group.
  Dose for BMI less than 35: 1.0 mg
  Dose for BMI greater than or equal to 35: 2.0 mg
  Other Names: Versed
Drug: Microcrystalline Cellulose — This will be used for the oral placebo. This capsule or a triazolam capsule will be administered depending on the randomized treatment group.
  Dose for BMI less than 35: 1 capsule
  Dose for BMI greater than or equal to 35: 2 capsule
  Other Names: Avicel
Drug: Sodium chloride 0.9% — This will be used for the intravenous placebo.This injection or midazolam will be administered depending on the randomized treatment group.
  Dose for BMI less than 35: volume to match volume of active intravenous medication
  Dose for BMI greater than or equal to 35: volume to match volume of active intravenous medication
  Other Names: Normal Saline

SUMMARY:
The purpose of this study is to evaluate patient satisfaction after eye surgery when given a capsule compared to an intravenous (IV) dose of sedation (calming medication).

Each subject will be given a capsule and an IV in the hospital before their procedure starts, however they will not know which one is the sedation route. Each subject will have their planned surgical procedure as previously discussed with their doctor. After the procedure is completed, the doctors will complete satisfaction surveys. The subject will also complete a satisfaction survey during their regularly scheduled visit the day after surgery. Once the subject completes this survey, their study participation will be complete.

The hypothesis is that there will be no difference in patient satisfaction when given a capsule in comparison to IV sedation. If the results of the study support this hypothesis, a capsule could be used in place of IV sedation. By using a capsule for ocular procedures, both patients and the medical practice would benefit: patient would be able to eat before their procedure, patient costs would be decreased, hospital costs would be reduced, and some of these procedures would be given the option to move to a procedure room (freeing up operating room time for other departments).

DETAILED DESCRIPTION:
The primary objective of this study is to compare patient satisfaction of oral triazolam to IV midazolam when administered for ocular procedures. Midazolam is an FDA-approved intravenous medication commonly used as a sedative for ocular procedures conducted in the operating room. This study will compare the use of triazolam, an FDA-approved oral sedative for the same types of ocular procedures, a purpose which has not fully been investigated. The benzodiazepine triazolam was chosen as the oral medication due to its similarity to midazolam. The similarities between midazolam and triazolam include similar half-life, risks, and patient experience.The medication doses were chosen from current SOC use based on weight. The lower dose for both medications are used for patients with a BMI less than 35 and the higher dose is used for patients with a BMI greater than or equal to 35.

This is the first double-blind, prospective clinical trial that will compare IV and oral sedation for multiple ocular sub-specialty procedures. The procedures to be investigated include: cataract, retina, cornea, and glaucoma surgical groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Ability to speak and read in English or Spanish or Haitian Creole
3. Subjects able to consent for themselves
4. Outpatient surgical plan for any of the following procedures:

   * Cataract surgery: cataracts
   * Retina: pars plana vitrectomy, pars plana vitrectomy with cataracts, epiretinal membrane peel, pars plana lensectomy, and/or endolaser, silicone oil removal
   * Cornea: descemet stripping endothelial keratopathy, cataracts with descemet stripping endothelial keratopathy, descemet membrane endothelial keratoplasty, cataracts with descemet membrane endothelial keratoplasty, conjunctival and/or corneal lesion excisions, pterygium
   * Glaucoma: ahmed valve, ahmed valve with cataracts,trabeculectomy, trabeculectomy with cataracts, baerveldt, baerveldt with cataracts, endocyclophotocoagulation, endocyclophotocoagulation with cataracts, istent, istent with cataracts, kahook, kahook with cataracts, cypass, cypass with cataracts

Exclusion Criteria:

1. Surgical plan which includes general anesthesia
2. Hypersensitivity or allergy to benzodiazepines
3. Women who are pregnant, have a positive pregnancy test on the day of surgery, refuse a pregnancy test, or are nursing
4. Previous delirium after anesthesia with a benzodiazepine
5. Subjects 70 years of age or older who fail the delirium pre-screening questionnaire as shown in Appendix Section 15.6
6. Currently experiencing the effects of drug/alcohol
7. Current oral/IV regimen of any medication inhibiting cytochrome P450 3A which includes ketoconazole, itraconazole, nefazodone, ritonavir, indinavir, nelavir, saquinavir, and lopinavir
8. Subjects already enrolled in this study for the fellow eye
9. Subjects enrolled in a clinical trial with an investigational drug within the past 3 months
10. Failed anesthesia clearance to receive a benzodiazepine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manju Subramanian, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ianchulev T, Litoff D, Ellinger D, Stiverson K, Packer M. Office-Based Cataract Surgery: Population Health Outcomes Study of More than 21 000 Cases in the United States. Ophthalmology. 2016 Apr;123(4):723-8. doi: 10.1016/j.ophtha.2015.12.020. Epub 2016 Jan 22. PMID 26804760
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Campbell J. Intravenous cannulation: potential complications. Prof Nurse. 1997 May;12(8 Suppl):S10-3. PMID 9180592
- [Background] Committee on Standards and Practice Parameters; Apfelbaum JL, Connis RT, Nickinovich DG; American Society of Anesthesiologists Task Force on Preanesthesia Evaluation; Pasternak LR, Arens JF, Caplan RA, Connis RT, Fleisher LA, Flowerdew R, Gold BS, Mayhew JF, Nickinovich DG, Rice LJ, Roizen MF, Twersky RS. Practice advisory for preanesthesia evaluation: an updated report by the American Society of Anesthesiologists Task Force on Preanesthesia Evaluation. Anesthesiology. 2012 Mar;116(3):522-38. doi: 10.1097/ALN.0b013e31823c1067. No abstract available. PMID 22273990
- [Result] Fung D, Cohen M, Stewart S, Davies A. Can the Iowa Satisfaction with Anesthesia Scale be used to measure patient satisfaction with cataract care under topical local anesthesia and monitored sedation at a community hospital? Anesth Analg. 2005 Jun;100(6):1637-1643. doi: 10.1213/01.ANE.0000154203.00434.23. PMID 15920188
- [Result] Erdurmus M, Aydin B, Usta B, Yagci R, Gozdemir M, Totan Y. Patient comfort and surgeon satisfaction during cataract surgery using topical anesthesia with or without dexmedetomidine sedation. Eur J Ophthalmol. 2008 May-Jun;18(3):361-7. doi: 10.1177/112067210801800308. PMID 18465717
- See also: Midazolam Drug Label Information — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=575d8bf0-7af7-427c-a231-966e2a5e070d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from October 26th, 2017 to November 30th, 2019 at the outpatient eye clinic, Ophthalmology Department, Boston Medical Center.
Pre-assignment Details: Out of 327 patients enrolled, 283 completed study participation and 44 patients did not complete study participation as they were dropped or withdrew from the study. 22 patients were dropped before randomization and 22 patients discontinued from study after randomization due to reasons seen in the participant flow table.
Groups:
- Retina Procedures: The following ocular procedures will fall under this arm of the study:
  * Pars plana vitrectomy (PPV)
  * PPV with cataracts, epiretinal membrane peel, pars plana lensectomy, and/or endolaser, silicone oil removal
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
- Cornea Procedures: The following ocular procedures will fall under this arm of the study:
  * Descemet Stripping Endothelial Keratoplasty (DSEK)
  * Cataracts with DSEK
  * Descemet Membrane Endothelial Keratoplasty (DMEK)
  * Cataracts with DMEK
  * Conjunctival and/or corneal lesion excisions
  * Pterygium
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
Period: Overall Study
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Started | 99 | 91 | 85 | 52
Completed | 85 | 84 | 70 | 44
Not Completed | 14 | 7 | 15 | 8
Not completed — Withdrawal by Subject | 5 | 2 | 4 | 2
Not completed — Ineligible on day of surgery | 7 | 2 | 0 | 3
Not completed — Study completed before surgical date | 2 | 1 | 8 | 1
Not completed — Transferred to other arm | 0 | 0 | 1 | 0
Not completed — Unable to obtain medication timely | 0 | 2 | 2 | 1
Not completed — Re-consented to participate | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The data displays information for participants that complete study participation.
Groups:
- Cataract Procedures: The following ocular procedures will fall under this arm of the study:
  • Cataracts
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Triazolam or microcrystalline cellulose oral placebo: Administered 30 minutes prior to surgery.
  Dose for BMI less than 35: 0.125 mg Dose for BMI greater than or equal to 35: 0.25 mg
  Midazolam or sodium chloride 0.9%: Administered 5 minutes prior to surgery Dose for BMI less than 35: 1.0 mg Dose for BMI greater than or equal to 35: 2.0 mg
- Retina Procedures: The following ocular procedures will fall under this arm of the study:
  * Pars plana vitrectomy
  * Pars plana vitrectomy with cataracts, epiretinal membrane peel, pars plana lensectomy, and/or endolaser, silicone oil removal
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Triazolam or microcrystalline cellulose oral placebo: Administered 30 minutes prior to surgery.
  Dose for BMI less than 35: 0.125 mg Dose for BMI greater than or equal to 35: 0.25 mg
  Midazolam or sodium chloride 0.9%: Administered 5 minutes prior to surgery Dose for BMI less than 35: 1.0 mg Dose for BMI greater than or equal to 35: 2.0 mg
- Cornea Procedures: The following ocular procedures will fall under this arm of the study:
  * Descemet Stripping Endothelial Keratoplasty (DSEK)
  * Cataracts with DSEK
  * Descemet Membrane Endothelial Keratoplasty(DMEK)
  * Cataracts with DMEK
  * Conjunctival and/or corneal lesion excisions
  * Pterygium
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% intravenous placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Triazolam or oral placebo: Administered 30 minutes prior to surgery Dose for BMI less than 35: 0.125 mg Dose for BMI greater than or equal to 35: 0.25 mg
  Midazolam or sodium chloride 0.9%: Administered 5 minutes prior to surgery Dose for BMI less than 35: 1.0 mg Dose for BMI greater than or equal to 35: 2.0 mg
- Glaucoma Procedures: The following ocular procedures will fall under this arm of the study:
  * Ahmed valve
  * Ahmed valve with cataracts
  * Trabeculectomy
  * Trabeculectomy with cataracts
  * Baerveldt
  * Baerveldt with cataracts
  * Endocyclophotocoagulation (ECP)
  * ECP with cataracts
  * Istent
  * Cataracts with istent
  * Kahook
  * Cataracts with kahook
  * Cypass
  * Cypass with cataracts
  Each subject will receive a capsule and an intravenous injection; however, they will not know which one is administering the sedation. Each patient will be randomized to one of the two groups listed below within this arm of the study:
  * Triazolam oral sedation with sodium chloride 0.9% IV placebo
  * Microcrystalline cellulose oral placebo with midazolam intravenous sedation
  Triazolam or placebo: Given 30 minutes prior to surgery Dose for BMI less than 35: 0.125 mg Dose for BMI greater than or equal to 35: 0.25 mg
  Midazolam or placebo: Given 5 minutes prior to surgery Dose for BMI less than 35: 1.
- Total: Total of all reporting groups
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures | Total
Number analyzed (Participants) | 85 | 84 | 70 | 44 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.59 (9.14) | 57.02 (12.65) | 49.96 (14.99) | 66.52 (11.32) | 59.67 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 23 | 20 | 124
  Male | 42 | 46 | 47 | 24 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 21 | 42 | 8 | 98
  Not Hispanic or Latino | 58 | 60 | 26 | 32 | 176
  Unknown or Not Reported | 0 | 3 | 2 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 34 | 28 | 19 | 28 | 109
  White | 22 | 25 | 9 | 2 | 58
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 29 | 29 | 41 | 13 | 112
Language [Count of Participants; unit: Participants]
  English | 51 | 56 | 25 | 26 | 158
  Spanish | 26 | 20 | 42 | 9 | 97
  Haitian Creole | 8 | 8 | 3 | 9 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.12 (6.44) | 29.86 (6.1) | 29.91 (5.48) | 29.6 (5.94) | 29.77 (5.94)

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Patient satisfaction will be determined by completion of a 12 question satisfaction survey. The responses to each question will be graded on a scale from 1 to 6: 1 being the least satisfied and 6 being the most satisfied. After all answers are graded for one survey, they will be averaged to give an overall survey grade on the 1 to 6 scale per patient. Higher mean scores are associated with higher levels of satisfaction.
Time Frame: The patient satisfaction survey was administered up to two days after surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Number analyzed (Participants) | 85 | 84 | 70 | 44
score on a scale | 5.37 (0.57) | 5.23 (0.72) | 5.37 (0.68) | 5.05 (0.87)
Statistical Analysis 1: Comparison: Cataract Procedures vs Retina Procedures vs Cornea Procedures vs Glaucoma Procedures; Testable hypothesis: Patient satisfaction mean will be non-inferior when given oral triazolam in comparison to IV midazolam during all basic cataracts, retina, cornea, and glaucoma ocular procedures. Null hypothesis: The null hypothesis is that the oral sedation group will have a primary endpoint mean equal to or less than that of the IV sedation group by the non-inferiority margin or more; Test type: Non-Inferiority — A non-inferiority margin of 0.5, will assure that, if non-inferiority is proven, the mean patient satisfaction with oral sedation will correspond to scores corresponding to satisfied or higher. A 0.5 margin to be considered clinically similar enough to declare non-inferiority because it allows for expected patient satisfaction variability, and demonstrates ample justification for providers to offer oral sedation as a safe alternative; p < 0.05, ANCOVA — As a sensitivity analysis, an ANCOVA model will be fit to the data adjusting for factors that are out of balance following randomization. The mean difference between the adjusted means will be calculated; If lower bound of the 90% two-sided Confidence Interval of mean difference is higher than -0.5, the oral sedation will be deemed non-inferior to IV

2. Secondary Outcome: Surgeon Satisfaction
Description: Surgeon satisfaction will be determined by completion of a 5 question satisfaction survey. The responses to each question will be graded on a scale from 1 to 6: 1 being the least satisfied and 6 being the most satisfied. After all answers are graded for one survey, they will be averaged to give an overall survey grade on the 1 to 6 scale per surgeon Higher mean scores are associated with higher levels of satisfaction.
Time Frame: The surgeon satisfaction survey will be administered immediately after the completion of the surgery. .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Number analyzed (Participants) | 85 | 84 | 70 | 44
score on a scale | 5.28 (0.97) | 5.57 (0.84) | 5.34 (0.95) | 4.6 (1.37)
Statistical Analysis 1: Comparison: Cataract Procedures vs Retina Procedures vs Cornea Procedures vs Glaucoma Procedures; Null hypothesis: Mean surgeon satisfaction score for oral triazolam will be statistically significant in comparison to mean surgeon satisfaction score for IV midazolam during all cataracts, retina, cornea, and glaucoma ocular procedures. Alternate hypothesis: Mean surgeon satisfaction score for oral triazolam will not be statistically significant in comparison to mean surgeon satisfaction score for IV midazolam during all cataracts, retina, cornea, and glaucoma ocular procedures; Test type: Non-Inferiority — A non-inferiority margin of 0.5, will assure that, if non-inferiority is proven, the mean patient satisfaction with oral sedation will correspond to scores corresponding to satisfied or higher. We determined a 0.5 margin to be considered clinically similar enough to declare non-inferiority because it allows for expected patient satisfaction variability, and demonstrates ample justification for providers to offer oral sedation as a safe alternative; p < 0.05, ANCOVA — Surgeon satisfaction score will be independently analyzed. Summary statistics including, means, standard deviations along with points estimates of the mean difference between the two groups and 90% Confidence Intervals; If lower bound of the 90% two-sided Confidence Interval of mean difference is higher than -0.5, oral sedation will be deemed non-inferior to IV

3. Secondary Outcome: Anesthesiologist/Certified Registered Nurse Anesthetist (CRNA) Satisfaction
Description: Anesthesiologist/CRNA satisfaction will be determined by completion of a 5 question satisfaction survey. The responses to each question will be graded on a scale from 1 to 6: 1 being the least satisfied and 6 being the most satisfied. After all answers are graded for one survey, they will be averaged to give an overall survey grade on the 1 to 6 scale per anesthesiologist/CRNA. Higher mean scores are associated with higher levels of satisfaction.
Time Frame: The anesthesiologist/CRNA satisfaction survey will be administered immediately after the completion of the surgical case.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Number analyzed (Participants) | 85 | 84 | 70 | 44
score on a scale | 5.16 (0.96) | 5.14 (0.94) | 5.33 (0.81) | 4.9 (0.96)
Statistical Analysis 1: Comparison: Cataract Procedures vs Retina Procedures vs Cornea Procedures vs Glaucoma Procedures; Null hypothesis: Mean anesthesiologist/CRNA satisfaction score for oral triazolam will be statistically significant in comparison to mean anesthesiologist/CRNA satisfaction score for IV midazolam during cataracts, retina, cornea, and glaucoma procedures. Alternate hypothesis:Mean anesthesiologist/CRNA satisfaction score for oral triazolam will not be statistically significant in comparison to mean satisfaction score for IV midazolam during cataracts, retina, cornea, and glaucoma procedures; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.05, ANCOVA — Anesthesiologist/CRNA satisfaction score will be independently analyzed. Summary statistics including, means, standard deviations along with points estimates of the mean difference between the two groups and 90% Confidence Intervals; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Number of Participants Requiring Additional Anesthesia Intervention
Description: The number of subjects in each arm that received additional anesthetic agents during the operative procedure after the initial sedation.
Time Frame: Information regarding additional anesthesia intervention will be collected within 2 days of completion of the subjects surgical procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Number analyzed (Participants) | 85 | 84 | 70 | 44
Participants | 11 | 8 | 11 | 16
Statistical Analysis 1: Comparison: Cataract Procedures vs Retina Procedures vs Cornea Procedures vs Glaucoma Procedures; Null hypothesis:The total additional anesthesia interventions for oral triazolam will be statistically significant in comparison to additional anesthesia interventions for IV midazolam during cataracts, retina, cornea, and glaucoma procedures. Alternate hypothesis:The total additional anesthesia interventions for oral triazolam will not be statistically significant in comparison to additional anesthesia interventions for IV midazolam during cataracts, retina, cornea, and glaucoma procedures; Test type: Other — Additional anesthesia intervention will be using summary statistics including, counts and proportions along with point's estimates of the proportion difference between the two groups and 90% Confidence Intervals; p < 0.05, t-test, 2 sided

5. Other Pre Specified Outcome: Surgical Complication Rates
Description: The number of subjects in each arm that experienced a complication during the operative procedure after the initial sedation.
Time Frame: Information regarding surgical complications will be collected within 2 days of completion of the subjects surgical procedure.
Population: Data was not available for one participant in the cornea arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
Number analyzed (Participants) | 85 | 84 | 69 | 44
Participants | 11 | 8 | 1 | 6
Statistical Analysis 1: Comparison: Cataract Procedures vs Retina Procedures vs Cornea Procedures vs Glaucoma Procedures; Null hypothesis: The total surgical complications for oral triazolam will be statistically significant in comparison to total surgical complications for IV midazolam during all cataracts, retina, cornea, and glaucoma ocular procedures. Alternate hypothesis: The total surgical complications for oral triazolam will not be statistically significant in comparison to total surgical complications for IV midazolam during all cataracts, retina, cornea, and glaucoma ocular procedures; Test type: Other — Surgical complications will be using summary statistics including, counts and proportions along with point's estimates of the proportion difference between the two groups and 90% Confidence Intervals; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were noted during the surgery and up to two days after the surgery when the patient satisfaction survey was administered.
Description: The same definition of adverse events and serious adverse events as clinicaltrials.gov. With the exception of hypertension, all other adverse events were not related to a particular organ system and occurred as a result of the surgical procedure.
Arm/Group | Cataract Procedures | Retina Procedures | Cornea Procedures | Glaucoma Procedures
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84 | 0/70 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/84 | 0/70 | 0/44
Other Adverse Events (participants affected / at risk) | 8/85 | 17/84 | 6/70 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cataract Procedures (N=85) | Retina Procedures (N=84) | Cornea Procedures (N=70) | Glaucoma Procedures (N=44)
In-patient Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient experienced pain and unease during surgery, and nausea, and malaise after surgery. The intervention was in-patient hospitalization. SAE was unexpected and the severity grade of SAE was 3. SAE was resolved on day of surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cataract Procedures (N=85) | Retina Procedures (N=84) | Cornea Procedures (N=70) | Glaucoma Procedures (N=44)
Pain During Surgery (Surgical and medical procedures) | 1 (1) | 15 (15) | 5 (5) | 3 (3) — The patient experienced pain and up to two days after surgery (in the eye, chest, back). The pain varied in severity and was self-reported by patients when the patient satisfaction survey was administered.
Nausea & Vomiting Post-surgery (Surgical and medical procedures) | 2 (2) | 7 (7) | 1 (1) | 1 (1) — The patient experienced nausea and vomiting after surgery. This was self-reported, varied in severity, and was recorded when the patient satisfaction survey was administered.
Headache & Dizziness (Surgical and medical procedures) | 3 (3) | 2 (2) | 3 (3) | 2 (2) — The patient experienced headache and/or dizziness after surgery. This was self-reported, varied in severity, and was recorded when the patient satisfaction survey was administered.
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The patient experienced hypertension after surgery. This was self-reported, varied in severity, and was recorded when the patient satisfaction survey was administered.
Anxiety (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The patient experienced anxiety before and during surgery. This was self-reported, varied in severity, and was recorded on the day of the surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03246724/Prot_SAP_000.pdf